CLINICAL TRIAL: NCT06233422
Title: Associations Between Actigraphy-Derived Sleep-Wake Patterns and Illness Trajectories and Treatment Response in Major Depressive Disorder
Brief Title: Longitudinal Ecological Study on Sleep-Wake Patterns in MDD Using Actigraphy
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Associate Professor, Chinese University of Hong Kong
Other Study IDs: PSY033
Record Dates: First submitted 2024-01-14; First posted 2024-01-31 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Depression; Sleep Disorders, Circadian Rhythm
Keywords: Actigraphy; Transdiagnostic Intervention; Depression; Rest-Activity Rhythm
MeSH Terms: conditions — Depression; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major Depressive Disorder (MDD) Group: MDD group will consist of 70 participants with MDD, aged between 18-65, with a Patient Health Questionnaire-9 (PHQ-9) score of at least 10; who are also experiencing at least 1 sleep or circadian problem in the past 3 months.
  Interventions: Other: No intervention involved
- Healthy Control Group: Healthy control group will consist of 70 healthy control participants, aged between 18-65, with a Patient Health Questionnaire-9 (PHQ-9) score of below 5, indicating minimal or no depressive symptoms.
  Interventions: Other: No intervention involved

INTERVENTIONS:
Other: No intervention involved — No intervention involved

SUMMARY:
The proposed study will include a longitudinal ecological study (Study 1) and a randomised controlled trial (Study 2). The aims will be to (1) identify the sleep-wake profiles in individuals with Major Depressive Disorder (MDD) through clustering; (2) examine the associations between sleep-wake features/profiles and the prognosis of MDD; and (3) investigate the anti-depressant effects of sleep- and circadian-targeted intervention in those with MDD and whether sleep-wake features/profiles may moderate the treatment outcomes.

In Study 1, a total of 140 participants comprising 70 participants with MDD and 70 age- and gender-matched healthy controls will be recruited. Sleep-wake patterns will be collected for 4 consecutive weeks using actigraphy devices and one-off self-report measures will be collected via an in-house smartphone application, PsyHub.

Study 1 and 2 will follow the CONSORT and STROBE guidelines, respectively. The current registration is only for Study 1 of the current research project.

ELIGIBILITY:
Inclusion Criteria for Healthy Control Group:

* Adults aged 18 to 65 years living in Hong Kong
* Being fluent and literate in Cantonese
* A Patient Health Questionnaire-9 (PHQ-9) score of below 5, indicating minimal or no depressive symptoms
* Accessibility to an Internet-enabled mobile device (iOS or Android operating system)
* Willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria for Healthy Control Group:

* Presence of any psychiatric disorder(s) as assessed by MINI
* Shift work, pregnancy, or work, family, or other commitments that interfere with regular sleep-wake patterns
* Presence of other untreated sleep disorders based on cut-off scores of individual sections in SLEEP-50.

We will not exclude those with current suicidal risks (i.e., non-fleeting intent or plan), which is a common symptom of MDD. However, if serious suicidal risk (i.e., PHQ-9 Item 9 score > 2) is identified, the participant will be referred to the PI (a clinical psychologist) for further assessment and professional mental health services if deemed necessary.

Inclusion Criteria for the Major Depressive Disorder (MDD) group:

* Adults aged 18-65 years living in Hong Kong
* Being fluent and literate in Cantonese
* A PHQ-9 score of at least 10, indicating a moderate level of depression.
* Meeting the DSM diagnostic criteria for current MDD according to the Mini International Neuropsychiatric Interview (MINI)
* Experiencing ≥ 1 sleep or circadian problem in the past 3 months according to the sleep and circadian problems checklist (i.e., time needed to fall asleep ≥ 30 minutes, wake after sleep onset ≥ 30 minutes, < 6-hour sleep per night or ≥ 9-hour sleep per night per 24-hour period, and falling asleep after 2:00 AM ≥ 3 nights per week; and variability in the sleep-wake schedule ≥ 2.78 hours within a week)
* Access to an Internet-enabled mobile device (iOS or Android operating system)
* Willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria for the Major Depressive Disorder (MDD) group:

* Severe medical or neurocognitive disorder(s) that make participation unsuitable based on the team's clinical experience
* Presence of other psychiatric disorders as assessed by MINI
* A history of electroconvulsive therapy (ECT)
* Current involvement in any psychological treatment programme that targets depression and/or sleep and circadian problems
* A change in the class or dose of any prescribed psychotropic drugs within 6 weeks before the baseline assessment
* Shift work, pregnancy, or work, family, or other commitments that interfere with regular sleep-wake patterns
* Presence of other untreated sleep disorders, including narcolepsy, obstructive sleep apnoea (OSA), and restless leg syndrome (RLS)/periodic leg movement disorder (PLMD) based on the cut-off scores of SLEEP-50 (narcolepsy ≥ 7; OSA ≥ 15; RLS/PLMD ≥ 7)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample, if recruitment in the community is insufficient, we will recruit participants from our collaborating outpatient clinics, non-governmental organizations, and community centers
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) | 1 at baseline, 4 weekly assessment across study 1, and 1 at the end of study 1
  A 9-item questionnaire used for screening, diagnosing, and monitoring the severity of depression, by scoring each item from "0" (not at all) to "3" (nearly everyday), total severity scale ranging from 0 to 27.
Change in Actigraphy (Actiwatch Spectrum Plus; USA Philips Respironics Inc.) - sleep onset latency (SOL) | 24-hour wear time for 4 consecutive weeks
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 4 consecutive weeks, SOL is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actiwatch Spectrum Plus; USA Philips Respironics Inc.) - wake after sleep onset (WASO) | 24-hour wear time for 4 consecutive weeks
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 4 consecutive weeks, WASO is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actiwatch Spectrum Plus; USA Philips Respironics Inc.) - total sleep time (TST) | 24-hour wear time for 4 consecutive weeks
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 4 consecutive weeks, TST is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actiwatch Spectrum Plus; USA Philips Respironics Inc.) - sleep efficiency (SE) | 24-hour wear time for 4 consecutive weeks
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 4 consecutive weeks, SE is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actiwatch Spectrum Plus; USA Philips Respironics Inc.) - fragmentation index (FI) | 24-hour wear time for 4 consecutive weeks
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 4 consecutive weeks, FI is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actiwatch Spectrum Plus; USA Philips Respironics Inc.) - time in bed (TIB) | 24-hour wear time for 4 consecutive weeks
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 4 consecutive weeks, TIB is one of the sleep parameters which will be measured by Actigraphy.
Change in Actigraphy (Actiwatch Spectrum Plus; USA Philips Respironics Inc.) - number of awakenings (NOA) | 24-hour wear time for 4 consecutive weeks
  Participants will be instructed to wear a wrist-worn actigraphy device to record their physiological patterns for 4 consecutive weeks, NOA is one of the sleep parameters which will be measured by Actigraphy.
Variability in sleep-wake variables using non-parametric approach - interdaily stability (IS) | 24-hour wear time for 4 consecutive weeks
  IS is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the non-parametric approach.
Variability in sleep-wake variables using non-parametric approach - intradaily variability (IV) | 24-hour wear time for 4 consecutive weeks
  IV is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the non-parametric approach.
Variability in sleep-wake variables using non-parametric approach - relative amplitude (RA) | 24-hour wear time for 4 consecutive weeks
  RA is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the non-parametric approach.
Variability in sleep-wake variables using non-parametric approach - the least active 5 hours (L5) | 24-hour wear time for 4 consecutive weeks
  L5 is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the non-parametric approach.
Variability in sleep-wake variables using non-parametric approach - the most active 10 hours (M10) | 24-hour wear time for 4 consecutive weeks
  M10 is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the non-parametric approach.
Variability in sleep-wake variables using extended cosinor approach - amplitude | 24-hour wear time for 4 consecutive weeks
  Rhythm height (amplitude) is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the extended cosinor approach. It tells the difference between the peak and nadir of the rhythm.
Variability in sleep-wake variables using extended cosinor approach - mesor | 24-hour wear time for 4 consecutive weeks
  Rhythm height (mesor) is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the extended cosinor approach. This tells the 24-hour adjusted mean rhythm activity,
Variability in sleep-wake variables using extended cosinor approach - acrophase | 24-hour wear time for 4 consecutive weeks
  Rhythm timing (acrophase) is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the extended cosinor approach. It tells the time of peak rhythm activity.
Variability in sleep-wake variables using extended cosinor approach - up-mesor | 24-hour wear time for 4 consecutive weeks
  Rhythm timing (up-mesor) is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the extended cosinor approach. This tells the activity initiation time.
Variability in sleep-wake variables using extended cosinor approach - down-mesor | 24-hour wear time for 4 consecutive weeks
  Rhythm timing (down-mesor) is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the extended cosinor approach. This tells the time of activity offset.
Variability in sleep-wake variables using extended cosinor approach - alpha | 24-hour wear time for 4 consecutive weeks
  Rhythm shape (alpha) is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the extended cosinor approach. This tells the width of the rhythm.
Variability in sleep-wake variables using extended cosinor approach - beta | 24-hour wear time for 4 consecutive weeks
  Rhythm shape (beta) is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the extended cosinor approach. It tells the steepness of the fitted curve.
Variability in sleep-wake variables using extended cosinor approach - pseudo F-statistic | 24-hour wear time for 4 consecutive weeks
  Rhythm robustness (pseudo F-statistic) is one of the sleep-wake variables which will be collected through Actigraphy, and quantified using the extended cosinor approach. This tells the goodness of extended cosine fit.

SECONDARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS) | 1 at baseline, and 1 at the end of study 1
  A 14-item scale measuring anxiety and depression in both hospital and community settings.
Change in Insomnia Severity Index (ISI) | 1 at baseline, and 1 at the end of study 1
  A 7-item scale used to assess the perceived severity of insomnia.
Change in Patient-Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD) and Sleep-Related Impairment (PROMIS-SRI) | 1 at baseline, 4 weekly assessment across study 1, and 1 at the end of study 1
  8-item scales to assess sleep and circadian functions.
Change in Multidimensional Fatigue Inventory (MFI) | 1 at baseline, and 1 at the end of study 1
  A 20-item scale used to assess five dimensions of fatigue.
Change in Short Form (6-Dimension) Health Survey (SF-6D) | 1 at baseline, and 1 at the end of study 1
  A health survey used for measuring the quality of life on six dimensions.
Change in Sheehan Disability Scale (SDS) | 1 at baseline, and 1 at the end of study 1
  A 5-item scale used to assess functional impairments in work/ school, social life, and family life.
Change in Core Consensus Standardized Sleep Diary | 4-week daily survey
  A 9-item scale used to record sleep time, wake time, perceived sleeping quality, and use of hypnotics.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong